CLINICAL TRIAL: NCT06210503
Title: The Comparison of Pericapsular Nerve Block and Fascia Iliaca Compartment Block in Children With Cerebral Palsy or Spina Bifida for Pain Management in Hip Surgery.
Brief Title: PENG Block in Comparison With FICB for Hip Reconstruction in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Novikova Veronika, Principal Investigator, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PENG vs FICB
Record Dates: First submitted 2023-12-21; First posted 2024-01-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Perioperative Analgesia; Hip Dislocation, Developmental
Keywords: Anesthesia local; nerve block; postoperative pain; hip dislocation; children
MeSH Terms: conditions — Developmental Dysplasia of the Hip; Pain, Postoperative; Hip Dislocation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG group (Active Comparator): The patient will undergo pericapsular nerve blockade with 0.5% ropivacaine based on 3 mg/kg ropivacaine using ultrasound scanning.
  Interventions: Procedure: Pericapcelar group nerve block
- FICB group (Active Comparator): The patient will undergo FICB with 0.5% ropivacaine based on 3 mg/kg ropivacaine using ultrasound scanning.
  Interventions: Procedure: Fascia iliaca compartment block

INTERVENTIONS:
Procedure: Pericapcelar group nerve block — In the supine position, a high-frequency linear sensor is placed in the anterior superior iliac spine and then aligned with the ramus of the pubis by rotating the probe counterclockwise approximately 45 degrees. The iliopsoas muscle and tendon, femoral artery, and pectineus muscle were observed in this view.The iliopsoas muscle and its tendon are visualized, as well as the vascular and nerve bundle: femoral artery, vein, and nerve. The needle is inserted laterally to medially in a planar approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the ramus pubis posteriorly. After negative aspiration, local anesthetic will be gradually injected aspirating every 3 mL.
  Arms: PENG group
Procedure: Fascia iliaca compartment block — In the supine position, a high-frequency linear sensor is placed in the inguinal fold. Scan starting lateral to the femoral artery and the nerve in the inguinal crease to identify the sartorius muscle, tracing the muscle to its origin to the anterior superior iliac spine. A shadow of the iliac crest bone and iliacus muscle will be visible, with the end point of injection being deep in the fascia iliaca and above the iliacus muscle at the lateral aspect of the iliacus muscle. After negative aspiration, local anesthetic will be gradually injected under the fascial plane, aspirating every 3 mL.
  Arms: FICB group

SUMMARY:
The goal of this clinical trial is to test the hypothesis that performing a Pericapsular nerve group (PENG) block allows for more effective analgesia in the perioperative period during reconstructive surgery on the hip in children with cerebral palsy and spina bifida compared with Fascia illiaca compartment block (FICB).

DETAILED DESCRIPTION:
The main question it aims to answer is: Is the PENG block an effective and safe method of pain relief for hip surgery in children? Participants will be randomized into two equal groups. The group who underwent US - guided PENG block, and the group who underwent US - guided FICB . In both groups we used 0.5% ropivacaine. The same postoperative analgesia regimen was applied by intravenous acetaminophen , oral ibuprofen . In case of ineffectiveness of the prescribed drugs, promedol was used intramuscularly. The postoperative consumption of promedol, time to first rescue analgesia, numerical pain score (NRS) (for children from 7 years old), FLACC score, measurements of A.N.I. monitor MDMS and the side effects will be recorded

ELIGIBILITY:
Inclusion Criteria:

* reconstructive surgery on the hip joint
* children with cerebral palsy/ spina bifida/organic brain injury
* age 3 - 18 years.

Exclusion Criteria:

* contraindications to the use of local anesthetics
* contraindications to performing an invasive procedure
* ASA > 3

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Opioids consumption | 24 hours
  Total dosage of opioids in postoperative period

SECONDARY OUTCOMES:
Time to rescue analgesia | 24 hours
  Time to first accepted of opioid analgesia
Pain level | 2, 6, 12, 24 hours after completing the block
  Assessing level of pain. Using pain scales. Face, Legs, Activity, Cry, Consolability (FLACC) scale for children from 3 to 7 years old. The scale is scored in a range of 0-10 with 0 representing no pain, and 10 representing maximal pain. The numeric rating scale (NRS) is a verbal or written determination of a pain level on a scale from 0 to 10, in which 0 represents no pain and 10 represents excruciating pain.
  Analgesia-nociception index (ANI). Using "ANI Monitor".
Intraoperative level of analgesia | Intraoperatively
  Analgesia-nociception index (ANI). Using "ANI Monitor".

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Petersburg State University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided